CLINICAL TRIAL: NCT02295397
Title: Integrated Approaches to Food Allergen and Allergy Risk Management
Acronym: iFAAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Cork University Hospital (Other); Charite University, Berlin, Germany (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Nebraska Lincoln (Other); Region Hovedstadens Apotek (Other Government); Servicio Madrileño de Salud, Madrid, Spain (Other); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: iFAAM
Record Dates: First submitted 2014-11-11; First posted 2014-11-20 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Food Allergy
Keywords: Food provocation; Matrix effect; ED05; Allergy; Proton Pump Inhibitor
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity | interventions — Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- food provocation (Experimental): open and placebo-controlled food challenges
  Interventions: Other: food

INTERVENTIONS:
Other: food — food provocation, skin testing, blood sampling

SUMMARY:
Patients with history of a food allergy to hazelnut, walnut or celeriac will undergo food provocation with a dose of the allergenic food to which 5% of the respective food allergic population (ED05) has been calculated to respond with allergic reactions (single shot study).

In patients with a hazelnut or peanut allergy a double-blind placebo controlled food challenge with cookies containing either placebo or hazelnut and peanut respectively will be performed to determine threshold levels eliciting an allergic reaction. The results for threshold levels determined by cookie matrix will be compared to the results gained from the EuroPrevall project (matrix comparison study).

In patients with a walnut allergy double-blind placebo controlled provocation with walnut will be combined with the intake of proton pump inhibitor (PPI) or with placebo to assess the impact of PPI on the threshold level and on the clinical manifestation.

DETAILED DESCRIPTION:
single shot study, matrix comparison and walnut/PPI study

1. detailed case history, blood sampling and prick testing with different foods will performed.
2. food provocation with a chocolate dessert meal containing either hazelnut, walnut or celeriac (ED05) will be performed (single shot study) in patients with a positive case history of an allergic reaction to either hazelnut, walnut or celeriac or with two meals containing either placebo or hazelnut and peanut respectively in hazelnut and peanut allergic patients or with three meals containing either placebo or walnut in walnut allergic patients.
3. in patients with a negative single shot challenge an open provocation with native hazelnut, walnut, celeriac will be performed unless the patients do not have had a positive previous food provocation with the respective food. In patients with a negative double-blind placebo-controlled food challenge an open provocation with hazelnut or peanut or walnut will be performed to confirm tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* For single shot study: history of a hazelnut, walnut, celeriac allergy due to an unequivocal accidental exposure with typical acute allergic reaction within the preceding 2 years and positive allergen-specific skin prick test/specific Immunoglobulin E or recent positive oral food challenge with hazel, walnut or celeriac within previous 2 years in children <16 years, but no time limit specified for adults
* For matrix comparison study: history of peanut or hazelnut allergy
* For walnut/PPI study: history of walnut allergy. The minimum age for this study is 18 years

Exclusion Criteria:

* Severe disease (heart, liver, kidney), acute febrile infection
* Intake of Ketotifen (past 2 weeks), corticosteroids (past 2 weeks), histamine-1-receptor blocker (past 3 days apart first generation past 7 days)
* Anaphylactic reaction (past 4 weeks)
* Uncontrolled bronchial asthma, forced expiratory volume < 70% predicted
* Pregnancy
* Acute infection or allergy
* Uncontrolled atopic dermatitis
* Chronic urticaria
* Mastocytosis
* Uncontrolled hypertension

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
numbers of patients reacting to ED05 in hazelnut, walnut, celeriac allergy | November 2014 to February 2017, up to 27 months

SECONDARY OUTCOMES:
numbers of patients reacting to a defined dose of peanut and hazelnut in titrated challenges | November 2014 to February 2017, up to 27 months
Change in the threshold dose of walnut that induces an allergic reaction after the intake of therapeutic doses of omeprazole Change in the severity of walnut allergy after the intake of therapeutic doses of omeprazole | February 2015 to February 2017, up to 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Clare Mills, Coordinator, Study Chair — University Manchester
Locations (1):
- Allergy Unit, Department of Dermatology, University Hospital, Zurich, Switzerland